CLINICAL TRIAL: NCT06535776
Title: Investigation of the Effect of Matrix Rhythm Therapy on Functional Status, Quality of Life, Respiratory Functions and Physical Performance in Axial Spondyloarthritis Patients
Brief Title: Effects of Matrix Rhythm Therapy in Axial Spondyloarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Ferruh Taşpınar, Study Director, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: matrix35
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Functional Status; Physical Performance

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Home-based exercise program will be explained to patients diagnosed with axSpA by a physiotherapist. All exercises will be repeated with the physiotherapist and explained until understood. Patients will be asked to perform these exercises on their own 3 non-consecutive days a week for 6 weeks. Patients will be called by the physiotherapist on each exercise day and their home exercises will be monitored and recorded in the exercise tracking chart created for each patient. In addition, the patients will be given an exercise follow-up chart and they will be asked to fill in the existing chart and submit it at the end of the 6-week training.
  Interventions: Other: Home-based Exercise
- Study group (Experimental): Individuals in this group will be taught home exercises face-to-face in a single session as in the home-based exercise group and will be asked to perform the exercises themselves at home for 3 non-consecutive days a week for 6 weeks. In this group, home exercises will be monitored by phone and recorded with an exercise tracking chart. In addition to home-based exercises, a total of 12 sessions of face-to-face matrix rhythm therapy will be performed, 2 non-consecutive days a week for 6 weeks. Matrix rhythm therapy applications will be applied by a specialist physiotherapist who has received training with the matrix rhythm therapy vibromassage device.
  Interventions: Other: Matrix Rhythm Therapy; Other: Home-based Exercise

INTERVENTIONS:
Other: Matrix Rhythm Therapy — Individuals in this group will be taught home exercises face-to-face in a single session as in the home-based exercise group and will be asked to perform the exercises themselves at home for 3 non-consecutive days a week for 6 weeks. In addition to home-based exercises, a total of 12 sessions of face-to-face matrix rhythm therapy will be performed, 2 non-consecutive days a week for 6 weeks. Matrix rhythm therapy applications will be applied by a specialist physiotherapist who has received training with the matrix rhythm therapy vibromassage device.
  Other Names: MRT
  Arms: Study group
Other: Home-based Exercise — Home-based exercise program will be explained to patients diagnosed with axSpA by a physiotherapist. All exercises will be repeated with the physiotherapist and explained until understood. Patients will be asked to perform these exercises on their own 3 non-consecutive days a week for 6 weeks. Patients will be called by the physiotherapist on each exercise day and their home exercises will be monitored and recorded in the exercise tracking chart created for each patient. In addition, the patients will be given an exercise follow-up chart and they will be asked to fill in the existing chart and submit it at the end of the 6-week training.
  Other Names: HBE

SUMMARY:
Axial spondyloarthritis (axSpA) is a chronic inflammatory rheumatic musculoskeletal disease affecting the axial skeleton. The most prominent symptom in patients with axial spondyloarthritis is morning stiffness and chronic low back pain. This is a chronic inflammatory disease group in which exercise and physiotherapy programs are recommended along with medical treatment. Considering the mechanism of action of matrix rhythm therapy, it was predicted that axial spondyloarthritis patients may show improvement.

DETAILED DESCRIPTION:
Axial spondyloarthritis (axSpA) is a chronic inflammatory rheumatic musculoskeletal disease affecting the axial skeleton. In addition to axial and musculoskeletal manifestations (arthritis, enthesitis, dactylitis), extramusculoskeletal manifestations (acute anterior uveitis, inflammatory bowel disease, psoriasis) are often present. In axSpA, the primary pathophysiology occurs in the entheses, the site of attachment of muscles to bones, and in the subchondral bone. In addition, secondary synovitis accompanies the pathology occurring in the enthesis. Mechanical stresses are very important in the onset and progression of axSpA. Axial inflammation causes bone destruction and plays an important role in the pathophysiology of axSpA.

The most common and frequently occurring symptom of axSpA is chronic (> 3 months) and almost daily chronic low back pain (CLBP) with morning stiffness. Pain and stiffness usually involve the lumbar region and buttocks, but any level of the spine can be affected. In addition, axial inflammation (synovitis and enthesitis) in axSpA causes irreversible structural damage and reduces spinal mobility. Spinal limitation is a late sign of axSpA.

Arthritis and enthesitis are the most common peripheral symptoms in axSpA and occur in approximately 30% of patients. Peripheral arthritis, which presents with edema and pain in the joints, is usually asymmetric monoarthritis/oligoarthritis and usually involves the lower extremities. Peripheral enthesitis usually presents with pain, stiffness and/or tenderness. Frequently, achilles enthesitis is seen in the lower extremities, but as axial enthesitis, it causes chest/back pain with synovitis of the axial joints. The combination of pharmacologic and non-pharmacologic methods in the treatment of axSpA has been shown to provide optimum benefit to patients. Pharmacologically, NSAIDs, tumor necrosis factor inhibitors, interleukin-17 inhibitors and Janus kinase inhibitors are preferred. In non-pharmacologic treatments, physiotherapy and exercise applications are recommended by the International Spondyloarthritis Society (ASAS-EULAR) with evidence grades 1a and 2b, respectively.

Exercise is the gold standard in the management of axSpA due to its proven benefits on disease outcomes independent of pharmacologic treatment. In the literature, studies conducted to evaluate the effects of exercise types (in-water exercises, group exercises, supervised individual exercises, aerobic exercises, pilates, tai-chi exercises, therapeutic exercises, proprioceptive exercises) on axSpA patients are frequently encountered. Due to the chronic nature of axSpA, continuity of treatment and time management, these exercises are modified and usually applied as home-based exercises. Home-based exercises are easily applicable and cost-effective, allowing patients to exercise while continuing their normal lives. In the literature, home-based exercise approaches have been shown to have positive effects on Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Bath Ankylosing Spondylitis Functional Index (BASFI), Bath Ankylosing Spondylitis Metrology Index (BASMI), scores, quality of life, pain and functional capacity in axSpA patients.

Exercise helps to regulate circulation, excrete metabolites and increase mitochondrial activity as a result of relaxation and contraction of muscles during activity. Some studies have shown pathological changes in the extracellular matrix of affected tissues in patients with axSpA. Successful treatment should focus on mobility of the extracellular matrix. Matrix metalloproteinase-mediated degradation of type II collagen, the main exacellular protein in cartilage, has been reported to be increased in patients with

ankylosing spondylitis (AS) and decreased with treatment. This is an important finding in diagnosis and prognosis. In order to correct this pathology in the matrix, supportive therapies that treat at the cellular level should be added together with exercise. It has been predicted that the effect of exercises will increase more with the reorganization of the extracellular matrix, restoration of its rhythm and regulation of circulation.

The Matrix Rhythm Therapy (MaRhyThe) vibromassage method for restoring the mobility and rhythm of the extracellular matrix was developed by Dr. Ulrich Randoll in Germany. This vibromassage device aims to reactivate cell metabolism by rhythmically stretching the deep tissue with its head. After micro stretching with the help of vibromassage, the tissues gain their unique natural vibration and the matrix rhythm improves. It has been reported that healthy muscles have vibrations between 8-12 Hz. and this is the same frequency as the alpha rhythm in the brain. However, if there is a pathology in the muscles, the vibration of the tissues is disturbed and the tissues move away from the alpha rhythm. It has even been reported that the rhythm of the tissues changes even during the day and metabolism is affected by this. In their study, Van Moorsel D examined the rhythms in skeletal muscles during the day and night by taking biopsy tissue from patients. They stated that the strong rhythms that change in biological clocks of individuals direct their oxidative metabolism. Disruption of these rhythms is associated with altered elasticity, plasticity and altered circulation at the cellular level.

There are studies in the literature using MaRhyThe in different populations. However, no studies have been found in patients with chronic and progressive axSpA affecting the extracellular matrix and peripheral tissues. AxSpA patients with axial skeletal involvement, which is frequently seen in the community, is a disease in which Matrix Rhythm Therapy can be applied. AxSpA is a chronic inflammatory disease group in which the use of exercise and supportive physiotherapy methods along with medical treatments is recommended in treatment guidelines. Therefore, in our study, it was decided to perform matrix rhythm therapy for the first time in AxSpA patients. Considering the mechanism of action of MaRhyThe, it is predicted to improve the effectiveness of exercise in patients with AxSpA by increasing the extracellular matrix fluid, excretion of metabolites and circulation. Therefore, our study was planned to examine the effect of Matrix Rhythm Therapy on functional status, quality of life, respiratory function and physical performance in patients with axSpA.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and over
* Individuals who can understand and respond to assessments
* Individuals followed with a diagnosis of axial spondyloarthritis for at least 6 months
* Individuals with a BASDAI score above 4

Exclusion Criteria:

* Individuals with unstable angina pectoris, uncompensated heart failure, myocardial infarction in the last month, which may pose a risk during exercise practices
* Individuals with uncontrolled diabetes, hypertension above 180/110 mmHg and/or severe neuropathy
* Individuals with diagnosed psychiatric illness
* Individuals with diagnosed severe cognitive impairment
* Individuals with severe dyspnea, cyanosis, hemoptysis at rest and/or minimal exertion
* Individuals with previous spinal injury and/or surgery
* Individuals with Psoriasis, Irritable Bowel Disease
* Individuals with pregnancy status/suspicion
* Patients with total ankylosis on direct radiograph or bamboo cane appearance on thoracolumbar radiograph

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-09-06 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | At baseline and after 6 weeks
  The BASDAI is a self-administered questionnaire consisting of six questions about the five main symptoms of fatigue, pain/swelling in the spine and joints, localized areas of tenderness and morning stiffness, measuring both severity and duration. Patients are asked to mark the extent to which they have experienced the relevant symptoms during the previous week. The first 5 questions are assessed using a visual analog scale with no markers on either end except for "not at all" and "very severe". For the amount of morning stiffness, the scale is graded in 15 minute intervals between 0-2 hours. The total score is calculated by averaging the total scale scores. A total score above 4 is considered active disease
Bath Ankylosing Spondylitis Functional Index (BASFI) | At baseline and after 6 weeks
  BASFI consists of 8 questions about functional activities in the last week and two questions assessing patients' ability to cope with daily life. Each question is answered on a 10 cm horizontal visual analog scale (VAS). There are no markings on the scale other than the words "easy" and "impossible" at both ends of the line to determine the direction of severity. The total score is calculated by averaging the ten questions, with higher scores indicating severe impairment.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | At baseline and after 6 weeks
  BASMI consists of 5 measurements: cervical rotation, tragus-wall distance, lateral flexion, modified schober distance and intermalleolar distance. Each measurement is scored between 0 (mild disease involvement) and 2 (severe disease involvement). Total BASMI score is between 0-10.
Ankylosing Spondylitis Quality of Life Questionnaire (ASYK) | At baseline and after 6 weeks
  The questionnaire consists of eighteen questions and each question is scored as yes-1 point and no-2 points. The total score ranges from 0-18, with a higher score indicating a worse quality of life.
Chest circumference measurement | At baseline and after 6 weeks
  Chest circumference measurement will be performed to evaluate chest expansion. In particular, in order to prevent contraction of the latissimus dorsi muscle and the associated misleading increase, the difference between maximum inspiration and expiration will be measured at the level of the 4th intercostal space with the patient's arms flexed in the frontal plane and the hands placed behind the head. A difference of less than 5 cm is considered significant for uptake
Pulmonary Function Test (PFT) | At baseline and after 6 weeks
  Pulmonary Function Test (PFT) is performed with a spirometer to evaluate lung volume and capacity. Lung functions of the patients will be evaluated with a spirometer (Cosmed Pony FX). As a result of the test, forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), FEV1/FVC values will be recorded.
Modified stoke ankylosing spondylitis spinal score (mSASSS) | At baseline and after 6 weeks
  Cervical and lumbar lateral radiographs, which are routinely ordered during the follow-up of the patients, will be evaluated according to the mSASSS system by the Rheumatology specialist of İzmir Buca Seyfi Demirsoy Training and Research Hospital. According to mSASSS, normal vertebrae are scored as 0, erosion/sclerosis/carring as 1, presence of syndesmophytes as 2, and ankylosis as 3 points. For cervical mSASSS, the upper and lower corners of all vertebrae between the lower corner of the C2 vertebra and the upper corner of the T1 vertebra will be evaluated. For lumbar mSASSS, the upper and lower corners of all vertebrae between the lower corner of the T12 vertebra and the upper corner of the sacrum will be evaluated. At the end of the assessment, the cervical mSASSS score, lumbar mSASSS score and total mSASSS score will be recorded.
Ankylosing Spondylitis Disease Activity Score (ASDAS) | At baseline and after 6 weeks
  ASDAS was developed in 2009 to assess disease activation. The ASDAS assessment consists of the second, third and sixth questions of the BASDAI, the patient's general self-assessment and the acute phase reactants CRP or ESR variables. The second, third and sixth questions of the BASDI are How would you describe the level of your neck, back, lower back and hip pain, How would you describe the level of your neck, back, lower back and hip pain and How long does your morning stiffness last after waking up? 0.12 x Back pain + 0.06 x Duration of morning stiffness + 0.11 x General assessment of the patient + 0.07 x Peripheral joint swelling/pain + 0.58 x Ln (CRP+1) to obtain the ASDASESH/CRP score and a score above 1.3 is considered active disease.
Sit-Bench Test | At baseline and after 6 weeks
  Hip and trunk flexibility will be assessed with the Sit-Bench Test. In this test, patients are placed in a long sitting position with their legs straight. The wall of the sit-stand board is placed on the soles of the feet and then the patient is asked to reach forward without bending the legs. After three reaches, the patient waits for two seconds and the distance between the fingertip of the hand and the board resting on the sole of the foot is recorded in +/- centimeters (cm).
Respiratory Muscle Strength | At baseline and after 6 weeks
  Respiratory muscle strength will be measured using MD Diagnostics Brand RP Check Respiratory Muscle Strength (Mip, Mep, Snip) Meter. Maximum inspiratory intraoral pressure and maximum expiratory intraoral pressure will be recorded.
6 Minute Walk Test (6MWT) | At baseline and after 6 weeks
  The 6DYT will be administered indoors in corridor lengths with smooth surfaces, at least 20 meters in length. In the test, with comfortable clothing and shoes suitable for walking, individuals will walk as quickly as possible at their own pace, stopping and using oxygen when necessary. Before and after the test, the heart rate, blood pressure and oxygen saturation (SpO2) of the individual will be measured; the degree of dyspnea according to the Borg scale and quadriceps fatigue will be questioned. At the end of the test, the reason and duration of rest, if any, will be recorded and the individual's six-minute walking distance will be determined in meters.
Chair Sit Up Test | At baseline and after 6 weeks
  A simple and quick test commonly used in the clinic to measure functional mobility.For the chair sit up test, the patient will sit in the center of a standard chair with their feet touching the floor. The patient will be asked to sit and stand in this position for 30 seconds without support and the total number of full sit-ups during this time will be recorded. Higher number of repetitions indicates better performance.
Timed Get Up and Go (SDG) Test | At baseline and after 6 weeks
  The SDM is a simple and rapid test widely used in the clinic that measures functional mobility of the lower limb, fall risk and performance. According to test scores <10sec = mobile, 10-20 s = usually independent > 30 sec = classified as restricted mobile For the SKY test, subjects will sit upright on a standard stool with their feet on the floor. With the command 'start', the patient will be asked to get up without holding on, walk towards an object 3 meters away, turn around, return to the chair and sit down. The time will start when the command is given and end when the person sits back in the chair. The elapsed time will be recorded with a stopwatch (sec).

CONTACTS AND LOCATIONS:
Overall Officials: Betül Taspinar, Prof.Dr., Principal Investigator — Izmir Democracy University; Onur Engin, Assist.Prof., Principal Investigator — Izmir Democracy University; Önay Gerçik, Assist.Prof., Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy Univercity, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navarro-Compan V, Sepriano A, El-Zorkany B, van der Heijde D. Axial spondyloarthritis. Ann Rheum Dis. 2021 Dec;80(12):1511-1521. doi: 10.1136/annrheumdis-2021-221035. Epub 2021 Oct 6. PMID 34615639
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/34615639/